CLINICAL TRIAL: NCT04216160
Title: Skin Acceptance and Efficacy Assessment of a Topical Product in Acne Treatment When Compared to a Placebo, Under Normal Use Conditions.
Brief Title: Skin Acceptance and Efficacy Assessment of a Topical Product in Acne Treatment When Compared to a Placebo.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: YUN NV (Industry)
Collaborators: Allergisa Pesquisa Dermato-Cosmetica LTDA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 074785-01/02-04-19-PRV03
Record Dates: First submitted 2019-12-26; First posted 2020-01-02 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Verum (Experimental): Patients with mild to moderate acne using ACN Cream
  Interventions: Other: ACN cream (YUN)
- Placebo (Experimental): Patients with mild to moderate acne using the placebo cream
  Interventions: Other: Placebo cream (YUN)

INTERVENTIONS:
Other: ACN cream (YUN) — Application of the facial cream ACN (YUN) twice a day, for 8 weeks +/- 2 days. Assessment before product use (T0), after 2, 4 and 8 weeks +/- 2 days of product use (T2w, T4w and T8w, respectively) and after 4 weeks +/- 2 days without product use (T12w).
  Other Names: Topical cream with live probiotic bacteria
  Arms: Verum
Other: Placebo cream (YUN) — Application of the facial placebo cream twice a day, for 8 weeks +/- 2 days. Assessment before product use (T0), after 2, 4 and 8 weeks +/- 2 days of product use (T2w, T4w and T8w, respectively) and after 4 weeks +/- 2 days without product use (T12w).
  Arms: Placebo

SUMMARY:
In this study the topical use of cream with live probiotic bacteria was evaluated for its efficacy in reducing acne symptoms and its effect on the skin microbiota on patients with acne vulgaris. Patients with mild to moderate acne used the probiotic cream for 8 weeks and clinical evaluation and microbiological sampling was done at start, 2, 4, 8 and 12 weeks (after 4 weeks without use of the product). Next-Generation Sequencing is used to analyze the skin microbiota of the patients.

DETAILED DESCRIPTION:
Probiotics are live micro-organisms which when administered in adequate amounts can exert a health benefit on the host. This health-promoting effects have been extensively studied in the gastrointestinal niche but it becomes more and more clear that other niches are also interesting for the potential of probiotics. Recent breakthroughs in 'next generation sequencing' (NGS) technologies are making it now possible to map the microbiota after DNA extraction, which is very interesting for bacteria that are not or difficult to cultivate. The research into the microbiota of the skin with such new NGS technologies shows that there is also an equilibrium in the skin composition of the microbiota and that there is a disturbance of the skin microbiota in acne. Acne vulgaris is known as a multifactorial condition, both hormonal triggers and environmental factors play a role. However, it is also known that Cutibacterium acnes and Staphylococcus spp. play an important role in the inflammation of the sebaceous gland follicles. Therefore, probiotic strains with antipathogenic activity against these bacteria and suitable for application to the skin are potentially able to restore the balance of the skin microbiota and reduce acne symptoms. The main objective of this study was to verify the skin acceptance and efficacy of the cream with live probiotic bacteria for acne treatment in comparison with a placebo. More specifically to evaluate the effect of the 'live' Lactobacillus species as 'active ingredient' in relation to acne symptoms and skin microbiome modulation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy skin in the test areas;
* Subjects willing and capable to follow the study rules and a fixed schedule;
* Ability of giving consent for participation in the study;
* Subjects with good health in general and good mental condition;
* Subjects who present at least 10 inflammatory lesions;
* Oily skin on the face (minimum sebumetry value 100µg/cm² on frontal area (mean: 3 measurements)).

Exclusion Criteria:

* Pregnancy or breastfeeding;
* Subjects who present severe acne;
* Subjects who present more than two nodular lesions;
* Subjects who changed their oral contraception method up to three months before the study beginning;
* Subjects who did acne hormonal treatment less than 6 months before the study;
* Subjects who did oral isotretinoïne treatment less than 1 month before the study;
* Subjects who did topical acne treatment less than 90 months before the study;
* Subjects who did aesthetic treatment less than 6 months before the study (like laser and peeling);
* Subjects who did treatment with antibiotics within the last 4 months;
* Simultaneous participation in different studies from external research institutes on the same test sites;
* Inadequate language proficiency (spoken and written);
* Participate in the study under the influence of alcohol and/or drugs as well as addiction;
* Severe psychological disease or intellectual disability of understanding the study;
* Severe disease (heart/circulatory/liver, kidney and lungs disease, severe diabetes mellitus) or chronic infections (hepatitis, HIV);
* Immune insufficiency;
* Current use of the following topical or systemic medications: corticosteroids, immunosuppressive and anti-histaminic drugs;
* Skin diseases: vitiligo, psoriasis, atopic dermatitis;
* Confirmed allergies to cosmetic components or previous responses of intolerance after the application of cosmetic products of the same category of the investigational products;
* Other diseases or medications that might directly interfere in the study or put the subject's health under risk.

Ages: 12 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2019-05-05 (Actual); Primary Completion 2019-11-28 (Actual); Study Completion 2020-02-11 (Actual)

PRIMARY OUTCOMES:
Change of inflammatory lesions compared to placebo. | baseline, 2, 4 and 8 weeks of product use and 4 weeks without product use (Total 12 weeks).
  The subjects were assessed by a trained technician in order to perform the acne lesions counting.
Change of inflammatory lesions compared to baseline. | baseline, 2, 4 and 8 weeks of product use and 4 weeks without product use (Total 12 weeks).
  The subjects were assessed by a trained technician in order to perform the acne lesions counting.
Overall tolerance of the treatment | Baseline to week 12
  Dermatological Assessment of Tolerance (DAT). On all visits, the dermatologist performed an assessment of the study subjects' faces according to a 5-point scale. The physician recorded in the subject's case report form possible discomforts sensation informed.

CONTACTS AND LOCATIONS:
Overall Officials: Mariane Mosca, Principal Investigator — Allergisa Pesquisa Dermato-Cosmética Ltda
Locations (1):
- Allergisa Pesquisa Dermato-Cosmética Ltda, Campinas, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No